CLINICAL TRIAL: NCT05581589
Title: A Pilot Single Arm Trial With Sacituzumab Govitecan as Neoadjuvant Therapy in Pts With Non-Urothelial Muscle Invasive Bladder Cancer
Brief Title: Sacituzumab Govitecan Before Radical Cystectomy for the Treatment of Non-Urothelial Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1122399; NCI-2022-04528 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10996 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-10-06; First posted 2022-10-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Muscle Invasive Bladder Carcinoma; Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Lymph Node Excision; Cystectomy; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sacituzumab govitecan) (Experimental): Patients receive sacituzumab govitecan IV over 3 hours on days 1 and 8 of each cycle. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Within 2-6 weeks after last dose, patients undergo radical cystectomy and pelvic lymph node dissection.
  Interventions: Procedure: Lymphadenectomy; Procedure: Radical Cystectomy; Biological: Sacituzumab Govitecan

INTERVENTIONS:
Procedure: Lymphadenectomy — Undergo pelvic lymph node dissection
  Other Names: excision of the lymph node; Lymph Node Dissection; Lymph Node Excision
Procedure: Radical Cystectomy — Undergo radical cystectomy
  Other Names: Complete Cystectomy
Biological: Sacituzumab Govitecan — Given IV
  Other Names: hRS7-SN38 Antibody Drug Conjugate; IMMU-132; RS7-SN38; Sacituzumab Govitecan-hziy; Trodelvy

SUMMARY:
This phase II trial tests whether sacituzumab govitecan given before radical cystectomy works in treating patients with non-urothelial bladder cancer. Sacituzumab govitecan contains a monoclonal antibody, called sacituzumab, linked to a chemotherapy drug, called govitecan. Sacituzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as TROP2 receptors, and delivers govitecan to kill them. Giving sacituzumab govitecan before radical cystectomy may make the surgery more effective in patients with muscle invasive bladder cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive sacituzumab govitecan intravenously (IV) over 3 hours on days 1 and 8 of each cycle. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Within 2-6 weeks after last dose, patients undergo radical cystectomy and pelvic lymph node dissection.

After completion of study treatment, patients are followed up at 1-3 months after radical cystectomy and then every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age on the day of signing informed consent. Participant (or legally acceptable representative if applicable) provides written informed consent for trial
* Participants must have either histologically or by clinical consensus (based on imaging and/or exam under anesthesia) confirmed diagnosis of muscle invasive bladder cancer (cT2-T4aN0-N1M0 or cT1-4aN1M0 clinical stage per American Joint Commission on Cancer [AJCC]). Patients with clinical node-positive (N1) stage are eligible provided the lymph node (LN) is confined to the true pelvis and is within the planned surgical LN dissection template; cN1 is defined as a lymph node with >= 15 mm short axis or biopsy-positive for carcinoma
* Must have clinical non-metastatic bladder cancer (M0) determined by cross-sectional Computed tomography (CT) chest, abdomen and pelvis (CAP) or magnetic resonance imaging (MRI)
* Review of pathology by local expert genitourinary (GU) pathologist is required. Any component (%) of non-conventional urothelial (variant histology) noted on transurethral resection of bladder tumour (TURBT) is allowed, for histologic types not listed below. However, for the variant histologic types listed below, the following parameters need to be met:

  * Squamous cell carcinoma / squamous cell features need to be pure or predominant (>= 1 variant histologic with total non-conventional urothelial component > 50%).
  * Adenocarcinoma / glandular features need to be pure or predominant (>= 1 variant histologic total non-conventional urothelial component > 50%).
  * Any % of neuroendocrine / small cell histology is excluded.
* Patients must be considered unfit for cisplatin based on the Galsky et al. criteria or refuse cisplatin despite adequate counseling in cisplatin-fit patients. Especially, for tumors containing squamous cell or glandular features, every effort should be made to discuss the benefit of neoadjuvant cisplatin-based chemotherapy shown in the S8710 trial
* Participants must be deemed eligible for radical cystectomy (RC) and pelvic lymph node dissection (PLND) by both urologist and medical oncologist
* TURBT that showed muscularis propria (or lamina propria for cT1N1 tumors) invasion should be within 12 weeks prior to beginning study therapy. Patients must have available tumor tissue from either initial or repeat TURBT, prior to starting study therapy. Archival and/or fresh tumor tissue sample of a tumor lesion (TURBT specimen) should be provided and must contain muscle invasive component, at least >= T2 tumor (for cT2 tumors), unless clinical stage is cT1N1M0 (in that case muscle invasive component is not necessary). Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory, preferably within 14 days from the date slides are cut if possible. Patient must be willing to provide tumor tissue for research. Research samples will not be used for unrelated studies
* A male participant must agree to use a contraception during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 180 days after the last dose of study treatment.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2. Patients with ECOG PS 2 may be permitted only after discussion with the trial primary investigator (PI) (Dr. Grivas). Evaluation of ECOG PS is to be performed within 7 days prior to the date of enrollment.
* Absolute neutrophil count (ANC) >= 1500/uL (within 10 days prior to the start of study treatment)
* Platelets >= 100 000/uL (within 10 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (within 10 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks prior to study drug treatment
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 30 ml/min (glomular filtration rate [GFR] can be used in place of creatinine clearance; 24-hour urine collection can be used for more accurate estimate as needed) (within 10 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 2.5 x ULN (within 10 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy (within 10 days prior to the start of study treatment)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy (within 10 days prior to the start of study treatment)
* Patients must agree to undergo curative intent surgery.

Exclusion Criteria:

* Patients with any % of neuroendocrine / small cell histology
* Patients considered to be medically unfit for SG, TURBT or radical cystectomy (per investigator discretion)
* Prior systemic anti-cancer therapy, including investigational agent/device within 4 weeks or prior radiation therapy within 2 weeks. Intravesical therapies are allowed without specified treatment interval
* Known locally advanced (unresectable, e.g. cT4b) or metastatic (cN2-3, M1) cancer on baseline radiographic imaging (CT or MRI) obtained within 28 days prior to registration
* Active infection requiring systemic antibiotic therapy at the time of trial initiation. Human immunodeficiency virus (HIV)-positive patients on active therapy are eligible as long as their viral load is undetectable and CD4 count is within normal parameters during the time of trial therapy initiation
* Known history of active hepatitis B (defined as hepatitis B surface antigen [HBsAg] detected or positive hepatitis B virus [HBV] polymerase chain reaction [PCR] test) or known active hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] detected) infection. Note: no testing for hepatitis B and hepatitis C is required if there is no clinical suspicion of such infection
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known personality, psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
* Patients may not have concurrent upper urinary tract (i.e., ureter, renal pelvis) invasive urothelial carcinoma. Patients with history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that have been definitively treated with at least one post-treatment disease assessment (i.e., cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible. Previously treated or concurrent non-invasive (Ta, Tis) urethra carcinoma is allowed, but history of or concurrent invasive urethra carcinoma is excluded
* Patients may not have another malignancy that could interfere with the evaluation of safety or efficacy of of SG. Patients with prior malignancy will be allowed without PI approval in the following circumstances:

  * Not currently active and completed therapy at least 2 years prior to the date of registration.
  * Non-invasive cancer, such as low risk cervical cancer or any carcinoma in situ.
  * Localized (early stage) cancer treated with curative intent (without evidence of recurrence and intent for further therapy), and in which no systemic chemotherapy was indicated (e.g., low/intermediate risk prostate cancer, non-melanoma skin cancer, etc.). Low/intermediate risk prostate cancer on active surveillance or watchful waiting is allowed. Other cancers not meeting these criteria must be discussed with trial PI (Dr. Grivas)
* Patients may not have undergone major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury =< 3 weeks prior to starting SG, or who have not recovered from side effects of such procedure or injury
* Have active (based on symptoms, endoscopic or biopsy findings) chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) at time of trial therapy initiation or history of GI perforation within 6 months of enrollment
* Patients may not have clinically significant cardiac diseases, including any of the following:

  * History or presence of serious uncontrolled ventricular arrhythmias.
  * Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, coronary artery bypass graft (CABG), New York Heart Association (NYHA) Class III or greater congestive heart failure (CHF) or left ventricular ejection fraction of < 40%, cerebrovascular accident (CVA), transient ischemic attack (TIA).
* Patients unwilling or unable to comply with the protocol or with known allergy to SG, its analogues, or excipients in the various formulations
* Patients may not participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial before radical cystectomy
* WOCBP with positive urine pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required for eligibility. Active lactation is exclusion
* History of allogeneic solid visceral organ transplant, Gilbert's disease, prior systemic irinotecan or topotecan or other topoisomerase-1 inhibitor, or concomitant medications that significantly interfere with ABCA1 transporter or UGT1A1 with no alternate option available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | At radical cystectomy (Radical cystectomy is expected to occur within 2-6 weeks after the last neoadjuvant trial therapy dose)
  pCR rate along with the 95% confidence interval (CI) based on the Clopper-Pearson method will be estimated.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) | At 2 years
  Kaplan-Meier (KM) method will be used to estimate RFS and corresponding 95% CIs, and the KM plots will be provided, when appropriate.
Overall survival (OS) | At 2 years
  KM method will be used to estimate OS and corresponding 95% CIs, and the KM plots will be provided, when appropriate.
Incidence of adverse events | Up to 2 years
  Assessed according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) in patients treated with SG.

CONTACTS AND LOCATIONS:
Overall Officials: Petros Grivas, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No